CLINICAL TRIAL: NCT05515705
Title: First-in-human Navigation Endoscopic Ultrasound (EUS) System Clinical Study
Acronym: APEUS-Nav1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of project funding and inclusion difficulties do not justify a request for extension.
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22-003
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2024-02

CONDITIONS: Pancreatic Disease
Keywords: Endoscopic ultrasound; EUS; Biliopancreatic; Pancreatic cancer; PDAC; EUS navigation; Education; Training; Learning curve; Quality indicators
MeSH Terms: conditions — Pancreatic Diseases; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- EUS-NS + (Experimental): EUS with the navigation system first on, then off
  Interventions: Device: EUS navigation system
- EUS-NS - (Experimental): EUS with the navigation system first off, then on
  Interventions: Device: EUS navigation system
- EUS group (No Intervention): EUS alone

INTERVENTIONS:
Device: EUS navigation system — Incorporation of the EUS navigation system to the EUS scope
  Arms: EUS-NS +; EUS-NS -

SUMMARY:
The implementation of Echo-endoscopy (or EUS for: Endoscopic UltraSound) is limited by the difficulty of obtaining quality EUS procedures, since the accuracy of the method relies on the endoscopist's abilities. Indeed, both cognitive and technical skills are required for endoscopic manipulation and image interpretation, as well as a thorough knowledge of intra-abdominal anatomy. The "EUS-GPS" system aims to assist the operator in understanding the orientation and location of the probe tip within the patient. For that, a Global Positioning System (GPS) for EUS procedures is intraoperatively provided, using a 3D-based model based on recorded preoperative data.

In this clinical investigation, the EUS GPS system is intended to help EUS operators to correctly navigate towards the pancreatic gland, perform a comprehensive assessment of the area of interest, and aid in the detection and identification of lesions.

DETAILED DESCRIPTION:
Since its emergence in the 1980s, endoscopic ultrasound (EUS) is considered as one of the most accurate tools for the evaluation of the pancreatic gland and other gastrointestinal (GI) disorders. Despite its utility, the practice of EUS is still far from being part of every endoscopy suite due to its high set-up cost and the relative scarcity of credentialed experts. EUS implementation worldwide has been limited by the difficulty of achieving quality EUS procedures, since the accuracy of the method relies on the endoscopist's abilities. Both cognitive and technical competencies are required for endoscopic manipulation and image interpretation, as well as extensive knowledge of intraabdominal anatomy.

The aim of the APEUS (Augmented Pancreatic Endoscopic UltraSound) project is to overcome these two main difficulties by providing a Global Positioning System (GPS)-like intraoperative navigation for EUS procedures, using a 3D-based model on registered preoperative data. The hypothesis is that, thanks to this tool, the procedures time would be shortened, and the pancreas and its lesions would be completely imaged. This would reduce the demand for experts guiding trainees and shorten the EUS learning curve.

This first-in-human clinical study will enable the assessment of safety and qualitative performance of the EUS-GPS solution. The primary objective is to evaluate the EUS navigation system's procedure duration compared to standard procedure times (patient group with the EUS-GPS system vs control group without).

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over the age of 18 years old
* Patient having a EUS procedure for pancreas study planned within the frame of his or her clinical care.
* Patient whom pre-operative imaging indicates one lesion with a good definition on the triphasic CT scan done within the 60 days prior to the EUS.
* Patient able to receive and understand information related to the study and give his or her written consent
* Patient affiliated to the French social security system

Exclusion Criteria:

* Patient unable to give informed consent
* Patient with altered anatomy of the upper digestive tract due to previous surgery
* Patient with known abnormal anatomy of the upper digestive tract
* Patient wearing a metal implantable device (pacemaker, etc.)
* Patient presenting, according to the investigator's judgment, a disease which may prevent participation in the procedures provided for by the study
* Patient with an ASA (American Society of Anesthesiologists) score >2
* Patient with multiple pancreatic lesions.
* Patient unable to tolerate general anaesthesia
* Patient with a body mass index (BMI) < 23 and > 40
* Patient with weight variations of >10% between the date on which the CT scan was performed and the date of the procedure.
* Pregnant or lactating patient
* Patient in exclusion period (determined by a previous or a current study)
* Patient under guardianship or trusteeship
* Patient under the protection of justice of deprives of liberty
* Patient in situation of emergency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the EUS navigation system's procedure duration compared to standard procedure times | 1 day
  Collect of peroperative duration for registration, insertion, navigation to cardia, navigation from the cardia to the pancreas, pancreas examination, therapeutic step and overall duration of the procedure (quantitative). Results will be compared between cases with (Groups EUS-NS) and without (Group EUS alone) use of the navigation system

SECONDARY OUTCOMES:
Assessment of the EUS navigation system in terms of reliability and safety | 1 day
  Rate of intraoperative undesirable events and of any event related to the tested system (probe breaking, software crashing, etc.)
Comparison of the EUS navigation system's procedure duration depending on the order the EUS-GPS is used | 1 day
  Collect of peroperative duration for registration, insertion, navigation to cardia, navigation from the cardia to the pancreas, pancreas examination, therapeutic step and overall duration of the procedure (quantitative). Results will be compared between cases with use of the navigation system first (Subgroup EUS-NS +) or in a second time (Subgroup EUS-NS -)
Assessment of the system's ease-of-use (integration in the standard-of-care workflow) compared to the standard procedure by the mean of a questionnaire | 1 day
  Questionnaire to assess the ease-of-use (integration in the standard-of-care workflow) of the EUS navigation system, filled by the EUS endoscopist (qualitative).
Assessment of the system's stressfulness compared to the standard procedure by the mean of a questionnaire | 1 day
  Questionnaire to assess the stressfulness of the EUS navigation system, filled by the EUS endoscopist (qualitative).
Collect adverse events, adverse device effects and device deficiencies | 1 month
  Collect adverse events, adverse device effects and device deficiencies during the procedure and up to 1 month after the EUS
Assessment of registration method by the mean of video recording analysis | 1 day
  A complete video recording of the procedure (endoscopic camera, ultrasound probe, pre-operative data real-time display and external camera) will be performed to assess the precision of the registration, using as anatomical points landmarks detectable in both CT and US images
Collection of EUS data | 1 day
  Videos of the EUS procedure for further use in Artificial Intelligence-driven EUS research projects will be collected if the patient specifically consents to it. Recorded material will include the electromagnetic (EM) coordinates provided by the sensor. EUS video data associated with EM coordinates will be used to build databases for AI-driven EUS research projects
Assessment of technological maturity and ergonomics | 1 day
  Questionnaire to evaluate the ergonomics and technological readiness, filled by the EUS endoscopist (qualitative).

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo SOSA VALENCIA, MD, Principal Investigator — IHU Strasbourg
Locations (1):
- Pôle Hépato-Digestif, NHC, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No